CLINICAL TRIAL: NCT07082218
Title: Multidimensional Sleep Health Intervention to Optimize Concussion Recovery: A Randomized Clinical Trial
Brief Title: Multidimensional Sleep Health Intervention to Optimize Concussion Recovery
Acronym: SCORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-2571
Record Dates: First submitted 2025-07-10; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Concussion (Diagnosis); Concussion, Mild Traumatic Brain Injury; Treatment; Sleep Health; Depression, Anxiety
Keywords: intervention; mild traumatic brain injury; sleep quality
MeSH Terms: conditions — Brain Concussion; Disease; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study will use a block stratified randomized clinical trial design. Our strata factor are the biological variable of sex and form of assessment (remote vs. in-person)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study principal investigator (PI) and the biostatistician will not know group assignments until after the primary analyses are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Sleep Intervention (Experimental): The intervention involves a structured intervention education session soon after enrollment, where participants receive tailored and personalized instructions for sleep health and quality, then complete daily adherence surveys, and receive follow-up support to address any barriers. The approach builds on prior work to address cognitive and emotional challenges commonly experienced by adolescents with concussion.
  Interventions: Behavioral: Sleep Intervention
- Standard-of-Care (No Intervention): Participants in the standard-of-care group will receive verbal and written sleep hygiene instructions at Visit 1, following established concussion management guidelines. These materials emphasize maintaining a consistent bedtime and reducing screen time before bed to support recovery. The approach reflects best practices informed by clinical recommendations for post-concussion care.

INTERVENTIONS:
Behavioral: Sleep Intervention — The investigators will randomly assign participants (adolescents with concussion) to a personalized sleep schedule and sleep health recommendation, based on a meeting with an administrator after enrollment and randomization. They will undergo testing prior to the intervention, after the intervention (2 weeks after the initial visit, intervention length=2 weeks), and 6 weeks after intervention completion.
  Arms: Individualized Sleep Intervention

SUMMARY:
Following adolescent concussion, poor sleep health is common and relates to the development of persisting post-concussion symptoms, and uninjured adolescents (independent of concussion) also commonly experience sleep insufficiency. Given the sparse guidance that exists for clinicians to provide evidence-based sleep health recommendations for adolescents with a concussion, the primary objectives of this prospective randomized clinical trial of adolescents with a recent concussion are to discover if a multidimensional and prescriptive sleep health intervention leads to: 1) faster symptom resolution time, better sleep quality, or longer sleep duration; and 2) improved sleep habits, mental health, or academic engagement, relative to standard-of-care post-concussion sleep health guidance. Findings from this research will provide the basis for more precise sleep health recommendations for adolescents who experience a concussion.

DETAILED DESCRIPTION:
Concussion is defined as a mild traumatic brain injury induced by biomechanical forces accompanied by an alteration in neurological status. Concussion recovery is complex, and many factors influence short- and long-term recovery outcomes. Among the deleterious effects observed after concussion, sleep-related problems are commonly reported and associated with increased risk of developing persisting post-concussion symptoms. Insufficient sleep is also commonly reported among uninjured adolescents, independent of concussion. In combination, adolescents with concussion are uniquely vulnerable to immediate and persisting sleep deficits. Currently prescribed sleep health recommendations for adolescents with a recent concussion remain vague, with limited evidence supporting intervention guidance. Given the documented relationship between post-concussion sleep problems and poor recovery outcomes, a multidimensional and prescriptive sleep health intervention initiated within the first month of a concussion may lead to improved patient outcomes. Using both patient-reported and objective (actigraphy) methods, our measurement approach will allow us to determine the efficacy of an innovative intervention to improve overall sleep health, concussion recovery, mental health, and academic engagement. The multidimensional sleep health intervention provides targeted and prescriptive recommendations for the patient and is developed from our existing pilot work. Specifically, the intervention addresses five areas with evidence to support post-concussion sleep deficits, including: 1) reduced time asleep, 2) inconsistent sleep/wake time, 3) more bed use for non-night-sleep purposes (e.g., napping), 4) excessive screen time before bed, and 5) night-time anxiety. Participants will be randomized to a multidimensional, prescriptive sleep health intervention or standard-of-care at Visit 1 (pre-intervention), undergo actigraphy monitoring and complete daily surveys for two weeks, return for re-assessment two weeks after Visit 1 (Visit 2, post-intervention), and 8 weeks after Visit 1 (Visit 3, persisting effects evaluation). Therefore, our objective is to discover if a multidimensional sleep health intervention among adolescents with a concussion (1) leads to faster symptom resolution time and better sleep quality and/or duration; and (2) affects persistent sleep habits, mental health, and academic engagement. We will use a two-group randomized clinical trial design (intervention, standard-of-care) with 3 assessments over an 8-week monitoring period. Our multidisciplinary investigative team, with expertise in concussion management, randomized clinical trials among adolescents with concussion, clinical trial design, and adolescent sleep behavior and psychology provides necessary experience to successfully complete this study. By challenging current sleep recommendations provided for adolescent patients with concussion, our project seeks to advance rehabilitation strategies for improved concussion management and overall improved health.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be symptomatic at the time of enrollment (Post-Concussion Symptom Inventory [PCSI] score ≥9)
* Diagnosed with a concussion by a healthcare provider using the American Congress of Rehabilitation Medicine diagnostic criteria
* 10-19 years of age (aligned with World Health Organization definition of 'adolescent')

Exclusion Criteria:

* History of treatment for pre-concussion sleep-related disorders

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Concussion symptom resolution time | Through study completion, an average of 8 weeks
  The day when symptoms are no longer experienced. As some may endorse symptoms independent of a concussion.

SECONDARY OUTCOMES:
Sleep duration | Through intervention completion, an average of two weeks
  Participants will wear a commercially available actigraphy device to quantify nightly sleep duration.
Sleep quality | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Self-reported measure of sleep quality perception completed via the Pittsburgh Sleep Quality Index. Scale=0-21, higher = worse sleep quality
Sleep disorders symptoms | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Sleep Disorders Inventory for Students; SDIS. T scores range from 0-90, and higher scores indicate more severe sleep disorder
Sleep behaviors | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Adolescent Sleep-Wake Scale; ASWS. Scores range from 28-168, with higher scores indicating better sleep quality.
Sleep onset and continuity | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Patient-Reported Outcomes Measurement Information System (PROMIS): Sleep Disturbance and Sleep-Related Impairment short forms. Scores are converted to T-scores, ranging from 35-75 with higher scores indicating more severe sleep problems
Sleep chronotype | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Morningness/Eveningness Scale for Children; MESC. Scores range from 10-50, with higher scores indicating a stronger morning preference and lower scores indicating a stronger evening preference.
Mental Health | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  PROMIS Global Pediatric Profiles 25, anxiety and depressive symptom domains. Scores are converted to T-scores with a range from 30-80, where higher scores indicate a more severe endorsement of anxiety and depressive symptoms.
Academic engagement | Baseline (Visit 1), Visit 2 (2 weeks after Visit 1), and Visit 3 (8 weeks after Visit 1)
  Identification with School Questionnaire; ISQ. Scores range from 16 to 80, with higher scores indicating a very high identification with school.

CONTACTS AND LOCATIONS:
Overall Officials: David R Howell, PhD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary deidentified outcome variables, demographics, and unblinded groups will be available based upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD and information will be available 6 months after the end of the trial (start date), for three years (end date)
Access Criteria: Researchers with adequate justification for reasonable as a part of other (e.g., meta-analytic) studies. Access to data will be granted via email communication.
URL: https://medschool.cuanschutz.edu/orthopedics/research/labs/howell-concussion-lab